CLINICAL TRIAL: NCT01021683
Title: The Relationship of Defeverscence and Itraconazole Plasma Level Using Sporanox IV as an Empiric Therapy in Immunocompromised Patients Who Have Been Treated With Sporanox Oral Solution as Prophylaxis
Brief Title: The Relationship of Defeverscence and Itraconazole Plasma Level Study in Immunocompromised Participants
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016597; ITR-KOR-5085; ITRFUN4049
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Hematologic Neoplasms; Neutropenia; Fever
Keywords: Hematological neoplasms; Neutropenia; Fever; Itraconazole; Sporanox; Antifungal prophylaxis; Defeverscence
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia; Fever | interventions — Itraconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood cultures
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Itraconazole: Participants who have been receiving itraconazole will be observed prospectively. Itraconazole will be administered as an infusion (a fluid or a medicine delivered into a vein by way of a needle) over one hour at the dose of 200 milligram (mg) per dose twice daily for 2 days, followed by 200 mg once daily for 12 days, followed by itraconazole oral solution at the dose of 200 mg per dose twice daily for 14 days until clinically significant neutropenia is recovered.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole will be administered as an infusion (a fluid or a medicine delivered into a vein by way of a needle) over one hour at the dose of 200 milligram (mg) per dose twice daily for 2 days, followed by 200 mg once daily for 12 days, followed by itraconazole oral solution at the dose of 200 mg per dose twice daily for 14 days until clinically significant neutropenia is recovered.

SUMMARY:
The purpose of this observational study is to investigate whether a sufficient concentration of itraconazole can influence disappearance of a fever (defeverscence) when intravenous (into the vein) itraconazole is administered for resolving unknown neutropenic fever of participants who are given itraconazole oral solution as a prophylaxis under general treatment conditions.

DETAILED DESCRIPTION:
This is a prospective (study following patients forward in time), open-label (all people know the identity of the intervention), multi-center (conducted in more than one center) observational study to examine the correlation between a sufficient blood concentration of itraconazole and disappearance of a fever (defeverscence) when itraconazole injection is administered for resolving unknown neutropenic fever of participants who are given itraconazole oral solution as a prophylaxis under general treatment conditions. The recommended dose of the drug will be 200 milligram (mg), which will be administered intravenously, twice daily for 2 days (a total of 4 doses) and then 200 mg once daily for 12 days. After the administration for a total of 14 days, itraconazole oral solution 200 mg (which is equivalent to 20 ml) twice daily will be continued for a total of 14 days until clinically significant neutropenia is resolved.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised participants with neutropenic fever who have been treated with itraconazole oral solution as prophylaxis
* Female participants who are postmenopausal or received contraceptive operation or refrain from sexual relations and women of childbearing potential should conduct an effective method of birth control (oral contraceptives, injections, intrauterine device, double barrier method, contraceptive patch and male partner's sterilization) before participation and during the study
* Male participants who will not have a baby within 2 months after the completion of itraconazole therapy

Exclusion Criteria:

* Fever due to documented deep-seated fungal infection at the entry into the study, but documented candidemia will be included
* Participants with kidney function related abnormalities with calculated creatinine clearance of 30 milliliter per minute (mL/min) or lower
* Aminotransferase level 5 times or higher of normal limit and total bilirubin level 5 milliliter per deciliter (mL/dL) or higher due to hepatic dysfunction
* Participants with dementia (mental decline) related to head injury and hypoxic brain injury
* Participants with mental illness which may interfere with cooperation in treatment and monitoring condition of the clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunocompromized participants with neutropenic fever who have been treated with itraconazole oral solution as prophylaxis and eligible for intravenous (into the vein) itraconazole in accordance with the local label.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole: Participants who had been receiving itraconazole were observed prospectively. Itraconazole was administered as an infusion (a fluid or a medicine delivered into a vein by way of a needle) over one hour at the dose of 200 milligram (mg) per dose twice daily for 2 days, followed by 200 mg once daily for 12 days, and then itraconazole oral solution at the dose of 200 mg per dose twice daily for 14 days until clinically significant neutropenia was recovered.
Period: Overall Study
Arm/Group | Itraconazole
Started | 203
Completed | 132
Not Completed | 71
Not completed — Lack of Efficacy | 12
Not completed — Recovery of neutrophil count | 51
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported only for intent-to-treat (ITT) population which included 150 participants.
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Plasma Level of Itraconazole at 1000 Nanogram Per Milliliter (ng/mL) or Higher After Administration of Study Treatment
Description: Percentage of participants who achieved more than or equal to 1000 ng/ml level after administration of study treatment were reported. Plasma level of itraconazole was defined as the sum of itraconazole concentration (IC) and hydroxyitraconazole concentration (HIC).
Time Frame: Day 5
Population: The intent-to-treat (ITT) population included the participants who satisfied the eligibility criteria, received the study drug at least once, and in whom the primary efficacy endpoint was measured at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Percentage of Participants | 68.0 [60.53 to 75.5]

2. Secondary Outcome: Percentage of Participants With Deferevescence After Administration of Study Treatment
Description: Defervescence was defined as fall of the body temperature below 38.0 degree Celsius (C) at least once after starting to receive the study treatment.
Time Frame: Day 0 up to Day 14
Population: The ITT population included the participants who satisfied the eligibility criteria, received the study drug at least once, and in whom the primary efficacy endpoint was measured at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Percentage of Participants | 87.3

3. Secondary Outcome: Mean Time to Defervescence in Participants Who Received the Study Treatment
Description: The mean time to defervescence was reported in participants who received the study treatment. Defervescence was defined as fall of the body temperature below 38.0 degree C at least once after starting to receive the study treatment.
Time Frame: Day 0 up to Day 14
Population: The ITT population included the participants who satisfied the eligibility criteria, received the study drug at least once, and in whom the primary efficacy endpoint was measured at least once. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Itraconazole
Number analyzed (Participants) | 131
Days | 3.14 (1.57) [2 to 13]

4. Secondary Outcome: Duration of Neutropenia
Description: The duration of neutropenia was reported. Neutropenia was defined as neutrophil count less than or equal to (<=) 500 cells per cubic millimeter (cells/mm^3), or neutrophil count <=1000 cells/mm^3 and anticipated to decrease to <=500 cells/mm^3 within several days.
Time Frame: Day 0 up to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Days | 2.64 (1.96)

5. Secondary Outcome: Absolute Neutrophil Count (ANC)
Description: The mean values for ANC based on blood tests performed on Day 0 (before starting the study treatment) constitute a Baseline measure for ANC.
Time Frame: Baseline (Day 0)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Itraconazole
Number analyzed (Participants) | 148
Cells/mm^3 | 56.26 (127.91)

6. Secondary Outcome: Percentage of Participants With Defervescence by Plasma Level of Itraconazole
Description: Defervescence was defined as fall of the body temperature below 38.0 degree C at least once after starting to receive the study treatment. Plasma level of itraconazole was defined as the sum of IC and HIC.
Time Frame: Day 5
Population: The ITT population included the participants who satisfied the eligibility criteria, received the study drug at least once, and in whom the primary efficacy endpoint was measured at least once. Here, 'n' signifies participants who were evaluable for this measure at given time points.
Measure: Number; unit: Percentage of Participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Percentage of Participants
  IC+HIC < 1000ng/mL (n=48) | 70.8
  IC+HIC >= 1000ng/mL (n=102) | 95.1

7. Secondary Outcome: Plasma Concentration of Itraconazole by Overall Success Rate (OSR) in Participants Who Received the Study Treatment
Description: Plasma level of itraconazole was defined as the sum of IC and HIC. The OSR was defined based on satisfaction of the following criteria: (1) participants if treated for baseline fungal infection, there was either eradication (removal of fungus in culture), or presumed eradication; no evidence in culture but appeared to be treated clinically, (2) absence of breakthrough fungal infection during the treatment and for 7 days after completing the treatment, (3) survival for 7 days after completing the treatment, (4) absence of early withdrawal due to adverse events or lack of efficacy, and (5) defervescence. The presence and absence of OS was reported.
Time Frame: Day 5
Population: The ITT population included the participants who satisfied the eligibility criteria, received the study drug at least once, and in whom the primary efficacy endpoint was measured at least once. Here, 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable for given category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Itraconazole
Number analyzed (Participants) | 134
ng/mL
  Presence of OS (n=95) | 2328.10 (1612.00)
  Absence of OS (n=39) | 1690.90 (1185.20)

8. Secondary Outcome: Percentage of Participants With Baseline Fungal Infection
Description: Blood cultures (a laboratory test on a sample of blood) were assessed to identify fungus. Percentage of participants with presence or absence of fungus before starting the study drug were calculated.
Time Frame: Baseline (Day 0)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 150
Percentage of Participants | 5.3 (1185.20)

9. Secondary Outcome: Plasma Concentration of Itraconazole by Breakthrough Fungal Infection
Description: Plasma level of itraconazole was defined as the sum of IC and HIC. A breakthrough fungal infection was defined as any fungal infection that was diagnosed more than (>) 3 days on or during therapy or within 7 days after completion of therapy. Blood cultures were assessed to identify fungus.
Time Frame: Day 5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Itraconazole
Number analyzed (Participants) | 134
ng/mL
  Presence of Breakthrough Fungal infection (n=128) | 2155.70 (1529.20)
  Absence of Breakthrough Fungal infection (n=6) | 1864.20 (1509.80)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 14
Arm/Group | Itraconazole
Serious Adverse Events (participants affected / at risk) | 28/203
Other Adverse Events (participants affected / at risk) | 49/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=203)
Bacterial sepsis (Infections and infestations) | 1
Cardiac arrest (Cardiac disorders) | 1
Disease progression (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Lung abscess (Infections and infestations) | 1
Multi-organ failure (General disorders) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia aspiration (Renal and urinary disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Sepsis (Infections and infestations) | 6
Septic shock (Infections and infestations) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=203)
Diarrhoea (Gastrointestinal disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Hemorroids (Gastrointestinal disorders) | 1
Lip disorder (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hepatic enzymes increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Pneumonia (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Oedema peripheral (General disorders) | 2
Asthenia (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Headache (Nervous system disorders) | 3
Depressed level of consciousness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arrhythmia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Disorientation (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot provide any trial related information to external parties without mutual agreement with the Sponsor. This is valid even after the contract is cancelled.